CLINICAL TRIAL: NCT03546426
Title: Pembrolizumab Plus Autologous Dendritic Cell Vaccine in Patients with PD-L1 Negative Advanced Mesothelioma Who Have Failed Prior Therapies
Acronym: MESOVAX
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST100.39
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Mesothelioma, Malignant; PD-L1 Negative; Advanced Cancer; Progressive Disease
Keywords: Mesothelioma, Malignant; PDL-1 negative; advanced disease; progressive disease
MeSH Terms: conditions — Mesothelioma, Malignant; Disease Progression | interventions — pembrolizumab; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- study treatment (Experimental): Pembrolizumab in combination with Autologous dendritic cells and Interleukin-2
  Interventions: Drug: Pembrolizumab; Biological: Autologous dendritic cells; Drug: Interleukin-2

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg IV q3w until disease progression, unacceptable toxicity or informed consent withdrawal, or for a maximum of 2 years
Biological: Autologous dendritic cells — Autologous dendritic cells (DC) loaded with autologous tumor homogenate, 10 x7 cells ID every 3 weeks for up to six doses
Drug: Interleukin-2 — 3 MU s.c. from day +2 to day +6 after each DC administration

SUMMARY:
Pembrolizumab plus autologous dendritic cell vaccine in patients with PD-L1 negative advanced mesothelioma who have failed prior therapies.This is an exploratory, single-arm, open-label, phase 1b clinical trial.

Patients will receive pembrolizumab 200 mg and autologous dendritic cell vaccine every 3 weeks for the first 6 cycles, followed by pembrolizumab 200 mg every 3 weeks until confirmed progression or for a maximum of 2 years (see Figure 1 Study Schema).

After each vaccine administration patients will receive IL-2 3 MU s.c. for 5 days, from day +2 to day +6.

DETAILED DESCRIPTION:
Pembrolizumab plus autologous dendritic cell vaccine in patients with PD-L1 negative advanced mesothelioma who have failed prior therapies.This is an exploratory, single-arm, open-label, phase 1b clinical trial.

The study will explore treatment safety and the ability to induce PD-L1 expression of the study treatment. Secondary objective will include clinical activity and immunological efficacy.

18 Patients will be enrolled . To ensure patients' protection and avoid unacceptable toxicity, a formal safety analysis will be conducted after six patients have been observed for at least 30 days after the third treatment cycle.

The study will be conducted on PD-L1 negative advanced mesothelioma patients with progressive disease after standard therapy. Previous therapies must have included an antifolate agent and a platinum compound.

Study treatment: Pembrolizumab 200 mg IV q3w until disease progression, unacceptable toxicity or informed consent withdrawal, or for a maximum of 2 years Autologous dendritic cells loaded with autologous tumor homogenate, 107 cells ID q3w for up to six doses Interleukin-2 3 MU s.c. from day +2 to day +6 after each DC administration.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed mesothelioma, with PD-L1 expression in less than 1% of cell in the screening tumor biopsy.
2. Progressive disease after at least one treatment line for advanced disease. Previous treatments must have included an antifolate agent and a platinum compound.
3. Patients must have recovered (grade 1 or less by CTCAE 4.0) from all the adverse events related to previous treatments.
4. The autologous surgical specimen needed for vaccine manufacturing must have been collected and sent to the Somatic Cell Therapy Lab of IRST IRCCS and must fulfil all the acceptance criteria prescribed by the GMP procedures.
5. Be willing and able to provide written informed consent/assent for the trial.
6. Be ≥ 18 years of age on day of signing informed consent.
7. Have measurable disease based on modified RECIST 1.0 for pleural mesothelioma or RECIST 1.1 for peritoneal mesothelioma.
8. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion (screening tumor biopsy). Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1.Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
9. Have a performance status of 0 or 1 on the ECOG Performance Scale.
10. Demonstrate adequate organ function as defined in Table 1; all screening labs should be performed within 10 days of treatment initiation.
11. Patients aged 70 years or older must have left ventricular ejection fraction not lower than 55% as assessed by echocardiography.
12. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. Female subjects of childbearing potential must be willing to use an adequate method of contraception . Contraception, for the course of the study through 120 days after the last dose of study medication.
14. Male subjects of childbearing potential must agree to use an adequate method of contraception - Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy > 10 mg prednisone equivalent or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Patients who have had chemotherapy, targeted small molecule therapy, or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events(i.e., ≤ Grade 1 or at baseline) due to agents administered more than 4 weeks earlier.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subjects received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Previous treatment with a cancer vaccine, or with agents targeting the PD-1/PD-L1 or PD-L2 axis.
8. Other known malignant neoplastic diseases in the patient's medical history with a disease-free interval of less than 5 years, except basal or squamous cell carcinoma of the skin and in situ carcinoma of the cervix uteri treated with radical surgery.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment, excepting for less than 10 mg prednisone equivalent. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has known history of, or any evidence of active, non-infectious pneumonitis or interstitial lung disease.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Any known history of or positivity of any serologic marker indicative of infection by Treponema pallidum, hepatitis B virus (HBsAg, HBsAb, HBcAB), hepatitis C virus (HCVAb, HCV RNA quantitative), human immunodeficiency virus (HIV), whether actual or previous. The sole positivity for antibodies against the HBsAg Ab (i.e. with all other HBV markers negative) is indicative of previous HBV vaccination and therefore is acceptable.
17. Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Safety as proportion of patients experiencing treatment-related adverse events | up to 90 days after end of study treatment
  The proportion of patients experiencing treatment-related grade 3-4 adverse events (AEs) according to NCI-CTCAE criteria, version 4.0.
PD-L1 expression induction by the treatment | up to 24 months
  Proportion of patients showing PD-L1 expression ≥ 1% of cells on post-treatment tumor samples.

SECONDARY OUTCOMES:
treatment activity | up to 24 months
  Clinical response by modified RECIST 1.0 for pleural mesothelioma and RECIST 1.1 criteria for peritoneal mesothelioma.
Immunological efficacy | up to 24 months
  Immunological activity will be evaluated by characterizing circulating immune response against universal and mesothelioma-associated tumor antigens by ELISPOT analysis and DTH skin test

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Guidoboni, MD, Study Chair — Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST)
Locations (1):
- Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC, Italy